CLINICAL TRIAL: NCT00934583
Title: Preventing Eating Disorders and Reducing Comorbidity
Brief Title: Testing an Internet-Based Intervention for Preventing Eating Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Craig Barr Taylor, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH081124 (NIH); R01MH081124 (NIH)
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Eating Disorders
Keywords: Bulimia Nervosa; Binge Eating; Binge-Eating Disorder
MeSH Terms: conditions — Feeding and Eating Disorders; Bulimia Nervosa; Bulimia; Binge-Eating Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Image and Mood (IaM) program (Experimental): Participants will participate in the IaM program.
  Interventions: Behavioral: Image and Mood (IaM) program
- Wait-list control (No Intervention): Participants will be placed on a wait list until after participants in the IaM group have completed all assessments. After that, these participants will be offered the option to complete the IaM program.

INTERVENTIONS:
Behavioral: Image and Mood (IaM) program — A 10-week Internet-based intervention focused on (1) identifying and challenging automatic thoughts in order to improve body image and reduce negative affect, (2) developing adaptive emotion and behavior regulation skills associated with preventing disordered eating and negative affect, and (3) teaching relapse prevention skills. The program includes an online discussion group moderated by a study clinician.
  Other Names: Student Bodies+
  Arms: Image and Mood (IaM) program

SUMMARY:
This study will examine the ability of an Internet-based program to prevent college-aged women from developing eating disorders.

DETAILED DESCRIPTION:
Approximately 2% to 4% of college-aged women suffer from eating disorders (EDs), and many more are at risk of developing them. A previous Internet-based intervention called Student Bodies (SB), which focused on body image concerns, was effective in reducing risk factors for EDs among college-aged women. However, the original SB program did not account for certain other risk factors, such as depression and compensatory behaviors like self-induced vomiting, over-exercising, or use of diuretics. Image and Mood (IaM) is an enhanced version of the SB program and takes into account depressive symptoms and the use of compensatory behaviors. This study will examine whether IaM will reduce ED risk factors in a large population of college women who are at high risk of developing EDs.

Participation in this study will last 10 weeks. Participants will be randomly assigned to either receive the IaM program or be placed on a wait list. The IaM program, which will be delivered through the Internet, will provide information about nutrition, exercise, body image, and coping skills-including examples and exercises. It will also include an online message board monitored by a study psychologist. Each week the IaM participants will monitor their behavior, keep a journal about their experiences, and answer self-report questionnaires. Assessments of eating disorder symptoms; weight and shape concerns; depressive symptoms; and incidence of substance abuse, anxiety, or depressive disorders will be completed post-treatment and at 1- and 1.5-month follow-ups. Those assigned to the wait list will complete these assessments and then receive the IaM program after the last follow-up.

ELIGIBILITY:
Inclusion Criteria for Primary Aim:

* Access to a computer with an Internet connection
* Weight Concerns Scale score greater than or equal to 47
* Presence of one additional risk factor, including a history of teasing, a history of depression, or low levels of compensatory behaviors (defined as less than four times per month)

Inclusion Criteria for Secondary Aim:

* Access to a computer with an Internet connection
* Weight Concerns Scale score greater than or equal to 47

Exclusion Criteria for Both Primary and Secondary Aims:

* Current diagnosis of an eating disorder
* Treated for an eating disorder within the past 6 months
* Currently receiving psychological treatment for an eating disorder or depressive disorder
* Started a new psychiatric medication within the past 2 months
* Exhibiting a level of psychopathology that would interfere with participation (e.g., acutely suicidal)

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 549 (Actual)
Dates: Start 2009-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Eating disorder diagnoses | Measured after 10 weeks, 1 year, and 1.5 years

SECONDARY OUTCOMES:
Weight Concerns Scale | Measured after 10 weeks, 1 year, and 1.5 years
Eating Disorder Examination Questionnaires (EDE-Q) | Measured after 10 weeks, 1 year, and 1.5 years
Depressive symptoms, as measured by the Beck Depression Inventory and Center for Epidemiologic Studies-Depression Scale | Measured after 10 weeks, 1 year, and 1.5 years
Combined incidence of substance abuse, alcohol abuse, anxiety disorders, and depressive disorders | Measured after 10 weeks, 1 year, and 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: C. Barr Taylor, MD, Principal Investigator — Stanford University; Denise Wilfley, PhD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Stanford, California
  - Washington University in St. Louis, St Louis, Missouri

REFERENCES:
- [Background] Taylor CB, Bryson S, Luce KH, Cunning D, Doyle AC, Abascal LB, Rockwell R, Dev P, Winzelberg AJ, Wilfley DE. Prevention of eating disorders in at-risk college-age women. Arch Gen Psychiatry. 2006 Aug;63(8):881-8. doi: 10.1001/archpsyc.63.8.881. PMID 16894064
- [Background] Taylor CB, Sharpe T, Shisslak C, Bryson S, Estes LS, Gray N, McKnight KM, Crago M, Kraemer HC, Killen JD. Factors associated with weight concerns in adolescent girls. Int J Eat Disord. 1998 Jul;24(1):31-42. doi: 10.1002/(sici)1098-108x(199807)24:13.0.co;2-1. PMID 9589309
- [Background] McKnight Investigators. Risk factors for the onset of eating disorders in adolescent girls: results of the McKnight longitudinal risk factor study. Am J Psychiatry. 2003 Feb;160(2):248-54. doi: 10.1176/ajp.160.2.248. PMID 12562570
- [Background] Wilfley DE, Welch RR, Stein RI, Spurrell EB, Cohen LR, Saelens BE, Dounchis JZ, Frank MA, Wiseman CV, Matt GE. A randomized comparison of group cognitive-behavioral therapy and group interpersonal psychotherapy for the treatment of overweight individuals with binge-eating disorder. Arch Gen Psychiatry. 2002 Aug;59(8):713-21. doi: 10.1001/archpsyc.59.8.713. PMID 12150647
- [Background] Wilfley DE, Cohen LR. Psychological treatment of bulimia nervosa and binge eating disorder. Psychopharmacol Bull. 1997;33(3):437-54. PMID 9550890
- [Background] Manwaring JL, Bryson SW, Goldschmidt AB, Winzelberg AJ, Luce KH, Cunning D, Wilfley DE, Taylor CB. Do adherence variables predict outcome in an online program for the prevention of eating disorders? J Consult Clin Psychol. 2008 Apr;76(2):341-6. doi: 10.1037/0022-006X.76.2.341. PMID 18377129
- [Background] Tanofsky-Kraff M, Wilfley DE, Young JF, Mufson L, Yanovski SZ, Glasofer DR, Salaita CG. Preventing excessive weight gain in adolescents: interpersonal psychotherapy for binge eating. Obesity (Silver Spring). 2007 Jun;15(6):1345-55. doi: 10.1038/oby.2007.162. PMID 17557971
- [Derived] Taylor CB, Kass AE, Trockel M, Cunning D, Weisman H, Bailey J, Sinton M, Aspen V, Schecthman K, Jacobi C, Wilfley DE. Reducing eating disorder onset in a very high risk sample with significant comorbid depression: A randomized controlled trial. J Consult Clin Psychol. 2016 May;84(5):402-14. doi: 10.1037/ccp0000077. Epub 2016 Jan 21. PMID 26795936